CLINICAL TRIAL: NCT05502081
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Antibodies Combination (Casirivimab and Imdevimab) Versus Standard Antiviral Therapy (Remdesivir and Favipravir) as Antiviral Agent Against Corona Virus 2 Infection in Hospitalized COVID-19 Patients
Brief Title: Clinical Study to Compare Efficacy and Safety of Casirivimab and Imdevimab Combination, Remdesivir and Favipravir in Hospitalized COVID-19 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed H Hassan, PharmD, Principal Investigator, Mansoura University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.21.11.1737; 35039/11/21 (Other: Tanta University)
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: COVID-19; Casirivimab & Imdevimab; Remdesivir; Favipravir
MeSH Terms: conditions — COVID-19 | interventions — casirivimab and imdevimab drug combination; remdesivir; favipiravir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- casirivimab and imdevimab (Experimental): casirivimab and imdevimab, vials 1.2 gm (1200 mg of combined antibodies) diluted in 250 ml 0.9% sodium chloride solution as single I.V infusion over 30-60 minutes.
  Interventions: Drug: Casirivimab and Imdevimab Drug Combination
- Remdesivir (Experimental): Remdesivir, vials Day1 (loading dose): 200 mg (two 100mg vials) diluted in 500ml 0.9% sodium chloride solution infused I.V over 60 minutes Day 2-5 or Day 2-10 (maintenance dose): 100 mg (one 100mg vial) in 250 ml 0.9% sodium chloride solution infused I.V over 30 minutes
  Interventions: Drug: Remdesivir
- Favipravir (Experimental): Favipravir, tablets Day 1 (loading dose): 1600 mg (8 tablets) or 1800 mg (9 tablets) orally or in Ryle tube / 12 hours Day 2-5 or day 2-10 (maintenance dose): 600 mg (3 tablets) or 800 mg (4 tablets) orally or in Ryle tube / 12 hours
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Casirivimab and Imdevimab Drug Combination — antiviral Monoclonal Antibodies
  Other Names: REGN-COV2
  Arms: casirivimab and imdevimab
Drug: Remdesivir — antiviral drug
  Other Names: Veklury
  Arms: Remdesivir
Drug: Favipiravir — antiviral drug
  Other Names: Avigan
  Arms: Favipravir

SUMMARY:
Introduction:

Corona Virus induced disease - 2019 (COVID-19) pandemic stimulates research works to find a solution to this crisis from starting 2020 year up to now. With ending of 2021 year, various advances in pharmacotherapy against COVID-19 have emerged.

Regarding antiviral therapy, Casirivimab and imdevimab antibody combination is a type of new immunotherapy against COVID-19. Standard antiviral therapy against COVID-19 includes Remdesivir and Favipravir.

Aim of Study:

1. To compare the efficacy of antibodies cocktail (casirivimab and imdevimab), Remdesivir and Favipravir in reducing 28-day mortality in hospitalized patients with moderate, severe or critical COVID19
2. To compare safety of antibodies cocktail (casirivimab and imdevimab), Remdesivir and Favipravir by monitoring hypersensitivity and infusion related reactions or other significant adverse effects

Patients and Population:

265 COVID-19 Polymerase Chain Reaction (PCR) confirmed patients with indication for antiviral therapy is included in this study and will be divided into 3 groups (1:2:2):

1. Group A: REGN3048-3051(Antibodies cocktail (casirivimab and imdevimab))
2. group B: Remdesivir
3. group C: Favipravir

Methods:

Study design is single blind non-Randomized Controlled Trial (non-RCT). The drugs of the study are owned by Mansoura University Hospital (MUH), and prescribed by chest diseases lectures of faculty of medicine-Mansoura University. The duration of study is about 6 months after ethical approval.

DETAILED DESCRIPTION:
I. INTRODUCTION

1.1. COVID-19 overview and classification

COVID-19 is an infectious viral disease caused by sever acute respiratory syndrome-corona virus 2 (SARS CoV-2) that has affected large number of people all over the world with high mortality rate. COVID-19 infection has been classified as:

1. Mild Illness: Individuals who have any of the various signs and symptoms of COVID-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and smell) but who do not have shortness of breath, dyspnea, or abnormal chest imaging.
2. Moderate Illness: Individuals who show evidence of lower respiratory disease during clinical assessment or imaging and who have an oxygen saturation (SpO2) ≥94% on room air at sea level.
3. Severe Illness: Individuals who have Saturation pressure of oxygen (SpO2) <94% on room air at sea level, a ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mm Hg, respiratory frequency >30 breaths/min, or lung infiltrates >50%.
4. Critical Illness: Individuals who have respiratory failure, septic shock, and/or multiple organ dysfunctions.

Covid-19 pandemic stimulates research works to find a solution to this crisis from starting 2020 year up to now. With ending of 2021 year, various advances in pharmacotherapy against COVID-19 have emerged.

1.2. Standard and controversial antivirals used in treatment of COVID-19 (Remdesivir and Favipravir)

Regarding antiviral drugs used in treatment of COVID-19, Remdesivir is a standard antiviral against COVID-19 and has been approved by Food and drug administration (FDA) for treatment of mild, moderate, sever and critical hospitalized COVID-19 patients. Other drugs have shown controversial antiviral activity include: favipravir, ivermectin, nitazoxanide, hydroxychloroquine, ribavirin. Favipravir became a standard antiviral which has been used for treatment of mild and moderate COVID-19 outpatients.

1.3. Advances in immunotherapy for treatment of COVID-19

Recently with the end of 2020, immunotherapy to target virus antigen has developed. Figure 1 shows two types of immunotherapy include active and passive immunotherapy. Active immunotherapy is to enhance body to produce antibodies against virus as by vaccination. Passive immunotherapy involves direct administration of prepared antibodies acting specifically against virus or administration of product containing antibodies like plasma.

There are three targets for these antibodies to work as antiviral including:

1. antibodies that prevent the virus attachment and entry
2. antibodies that inhibit the virus replication and transcription
3. antibodies that hinder various steps of the immune system response Table 1 includes various types of antibodies under investigation for treatment of COVID-19 and their targets.

1.4. Casirivimab and Imdevimab as antibodies cocktail against COVID-19

In the present study, the point of research is antibodies cocktail including REGN3048-3051(casirivimab and imdevimab).REGN3048 and REGN3051 are human monoclonal antibodies targeting the spike glycoprotein on surface of viral particles thereby preventing viral entry into human cells through the angiotensin-converting enzyme 2(ACE2) receptor, and have shown promising antiviral activity and need for further investigation to prove their benefit in COVID patients.

Previous study on REGN3048-3051 has mentioned that both efficacy and safety of this antibodies cocktail are proved in COVID-19 outpatients treatment in both low (2.4 g of REGN-COV2), or high (8.0 g of REGN-COV2) dose when compared to placebo, Efficacy is measured as

1. Virologic Efficacy Time-weighted average change from baseline in viral load through day 7 (log10 scale) in patient.
2. Clinical Efficacy Percentage of patients with one or more medically attended visits and Symptoms offset at day 7

Safety is measured as Percentage of treated patients who experience infusion related and hypersensitivity reactions and incidence of any serious and unexpected adverse effect.

This previous study concluded that efficacy is greater and more obvious in seronegative outpatients (whose immune response is not developed yet to produce antibodies against virus) and with high baseline viral load outpatients.

Now, data is available for these new antibodies cocktails. The U.S. FDA has allowed an Emergency Use Authorization (EUA) for casirivimab and imdevimab combination in the treatment and post-exposure prophylaxis of mild and moderate COVID-19 in adults and pediatric outpatients (more than12 years of age and not less than 40 kg) with positive PCR results of direct SARS-CoV-2 viral testing, and who are at high risk for progression to severe COVID-19 requiring hospitalization or causing death..

In contrast, REGN3048 and REGN3051 are still not authorized for use in patients:

* who are hospitalized due to COVID-19, OR
* who require oxygen therapy due to COVID-19, OR
* who require an increase in baseline oxygen flow rate due to COVID-19 in those on chronic oxygen therapy due to underlying non-COVID-19 related comorbidity(FDA, 2021).

Now, casirivimab and imdevimab are approved investigational antibodies, Serious and unexpected adverse effects can occur that not previously reported with their use.

Confirmed adverse effects include hypersensitivity and infusion related reactions and the study have showed that there is no difference in safety profile between intravenous (I.V) infusion and subcutaneous (S.C) injection. Data about use during pregnancy and breastfeeding mother is insufficient yet. Also, Data not support any dosage adjustment in hepatic and renal patients.

This antibody combination follows linear pharmacokinetics after its single intravenous doses with half-life of about 25 to 37 days for both antibodies. Regarding elimination, this combination is not metabolized by liver cytochrome enzymes ,and not excreted by kidneys.

Limitations of the previous study performed on antibody cocktail include:

1. short duration of follow up
2. not used much clinical relevant outcomes like mortality rate
3. Not studied the long term effect of antiviral efficacy in lowering viral load on inflammatory markers.
4. Study performed on non-hospitalized patients only and not included hospitalized patients (trial is done only on outpatients and not inpatients)

II. AIM OF THE STUDY:

1. To evaluate the efficacy of antibodies cocktail (casirivimab and imdevimab) compared to standard antiviral therapy in reducing 28-day mortality in hospitalized patients with moderate, severe or critical COVID19
2. To evaluate safety of antibodies cocktail (casirivimab and imdevimab) compared to standard antiviral therapy by monitoring of hypersensitivity and infusion related reactions or other significant adverse effects

III. PATIENTS AND POPULATION

265 COVID-19 PCR confirmed patients with indication for antiviral therapy is included in this study and will be randomized (2:1:1) into 3 groups

1. Group A: REGN3048-3051(Antibodies cocktail (casirivimab and imdevimab) )
2. group B: Remdesivir
3. group C: Favipravir

Population in this study are patients hospitalized in isolation hospital-Mansoura university.

A computer file containing a written informed consent from included patients will be provided. Paper will not be a tool for providing agreement by patients or their relatives to avoid transmission of infection.

IV. INTERVENTIONS

Population included in this study will be assigned into 3 groups with 1:2:2 ratios to receive either antibodies cocktail or standard antiviral therapy (remdesvir, favipravir).

Group A patients will receive REGN3048-3051(Antibodies cocktail (casirivimab and imdevimab) ) in low-dose regimen 1.2 gm (1200 mg of combined antibodies) diluted in 250 ml 0.9% sodium chloride solution as single I.V infusion over 30-60 minutes.

Group B patients will receive Remdesivir :

Day1 (loading dose): 200 mg (two 100mg vials) diluted in 500ml 0.9% sodium chloride solution infused I.V over 60 minutes Day 2-5 or Day 2-10 (maintenance dose): 100 mg (one 100mg vial) in 250 ml 0.9% sodium chloride solution infused I.V over 30 minutes

Group C patients will receive Favipravir :

Day 1 (loading dose): 1600 mg (8 tablets) or 1800 mg (9 tablets) orally or in Ryle tube / 12 hours Day 2-5 or day 2-10 (maintenance dose): 600 mg (3 tablets) or 800 mg (4 tablets) orally or in Ryle tube / 12 hours

Patients will be received standard of care by Physicians, Clinical pharmacist , Nurses and as guided by Egyptian COVID-19 treatment protocol.

V. METHOD

The type of this study is single blind non-RCT and is considered a Phase IV Clinical trial (post-marketing study) to report efficacy and safety of new medicine.

We use PubMed search tool to find clinical studies that performed to test efficacy and safety of developed immunotherapy in treatment of COVID-19 with about 4,000 results with focusing on antibodies developed as antiviral against COVID-19 obtaining only 70 results from which REGN-COV2, a Neutralizing Antibody Cocktail is selected with its only one clinical study up to now (REGN-COV2, a Neutralizing Antibody Cocktail, in Outpatients with Covid-19) which is published in New England Journal of Medicine on January 21, 2021.

Another resource used to obtain data is Fact Sheet for Health Care Providers- EUA OF casirivimab and imdevimab which provides clinical data about the use of this antibodies cocktail. Endnote citation software is used for citation of references.

ELIGIBILITY:
Inclusion Criteria:

1. age more than 12 years old.
2. weight not less than 40 kg.
3. Moderate, sever or critical COVID-19 disease as defined by WHO.
4. PCR- confirmed patients to be Positive before inclusion.

Exclusion Criteria:

1. history of hypersensitivity or infusion related reactions after administration of monoclonal antibodies.
2. prior use of standard antiviral therapy (remedsvir or favipravir).
3. Current use of controversial antiviral therapy (hydroxychloroquine, ivermectin, nitazoxanide, oseltemavir, acyclovir, ribavirine, lopinvir/rotinvir, sofosfbuvir, decltasevir, semipirvir, azithromycin).
4. patients expected to die within 48 hours.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shar K Hegazy, prof, Study Director — Tanta Unversity
Locations (1):
- El-gomhoria St, Al Mansurah, El-dkhalia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After the end and publication of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the end and publication of the study
Access Criteria: all will be accessiable

REFERENCES:
- [Background] Okonji EF, Okonji OC, Mukumbang FC, Van Wyk B. Understanding varying COVID-19 mortality rates reported in Africa compared to Europe, Americas and Asia. Trop Med Int Health. 2021 Jul;26(7):716-719. doi: 10.1111/tmi.13575. Epub 2021 May 1. PMID 33733568
- [Background] COVID-19 Treatment Guidelines Panel. Coronavirus Disease 2019 (COVID-19) Treatment Guidelines [updated September 29, 2021. Available from: https://www.covid19treatmentguidelines.nih.gov.
- [Background] Umakanthan S, Chattu VK, Ranade AV, Das D, Basavarajegowda A, Bukelo M. A rapid review of recent advances in diagnosis, treatment and vaccination for COVID-19. AIMS Public Health. 2021 Feb 1;8(1):137-153. doi: 10.3934/publichealth.2021011. eCollection 2021. PMID 33575413
- [Background] Aleem A, Kothadia JP. Remdesivir. StatPearls. Treasure Island (FL): StatPearls Publishing Copyright © 2021, StatPearls Publishing LLC.; 2021
- [Background] de Almeida SMV, Santos Soares JC, Dos Santos KL, Alves JEF, Ribeiro AG, Jacob ITT, da Silva Ferreira CJ, Dos Santos JC, de Oliveira JF, de Carvalho Junior LB, de Lima MDCA. COVID-19 therapy: What weapons do we bring into battle? Bioorg Med Chem. 2020 Dec 1;28(23):115757. doi: 10.1016/j.bmc.2020.115757. Epub 2020 Sep 10. PMID 32992245
- [Background] Owji H, Negahdaripour M, Hajighahramani N. Immunotherapeutic approaches to curtail COVID-19. Int Immunopharmacol. 2020 Nov;88:106924. doi: 10.1016/j.intimp.2020.106924. Epub 2020 Aug 21. PMID 32877828
- [Background] Baum A, Fulton BO, Wloga E, Copin R, Pascal KE, Russo V, Giordano S, Lanza K, Negron N, Ni M, Wei Y, Atwal GS, Murphy AJ, Stahl N, Yancopoulos GD, Kyratsous CA. Antibody cocktail to SARS-CoV-2 spike protein prevents rapid mutational escape seen with individual antibodies. Science. 2020 Aug 21;369(6506):1014-1018. doi: 10.1126/science.abd0831. Epub 2020 Jun 15. PMID 32540904
- [Background] Hansen J, Baum A, Pascal KE, Russo V, Giordano S, Wloga E, Fulton BO, Yan Y, Koon K, Patel K, Chung KM, Hermann A, Ullman E, Cruz J, Rafique A, Huang T, Fairhurst J, Libertiny C, Malbec M, Lee WY, Welsh R, Farr G, Pennington S, Deshpande D, Cheng J, Watty A, Bouffard P, Babb R, Levenkova N, Chen C, Zhang B, Romero Hernandez A, Saotome K, Zhou Y, Franklin M, Sivapalasingam S, Lye DC, Weston S, Logue J, Haupt R, Frieman M, Chen G, Olson W, Murphy AJ, Stahl N, Yancopoulos GD, Kyratsous CA. Studies in humanized mice and convalescent humans yield a SARS-CoV-2 antibody cocktail. Science. 2020 Aug 21;369(6506):1010-1014. doi: 10.1126/science.abd0827. Epub 2020 Jun 15. PMID 32540901
- [Background] Weinreich DM, Sivapalasingam S, Norton T, Ali S, Gao H, Bhore R, Musser BJ, Soo Y, Rofail D, Im J, Perry C, Pan C, Hosain R, Mahmood A, Davis JD, Turner KC, Hooper AT, Hamilton JD, Baum A, Kyratsous CA, Kim Y, Cook A, Kampman W, Kohli A, Sachdeva Y, Graber X, Kowal B, DiCioccio T, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD; Trial Investigators. REGN-COV2, a Neutralizing Antibody Cocktail, in Outpatients with Covid-19. N Engl J Med. 2021 Jan 21;384(3):238-251. doi: 10.1056/NEJMoa2035002. Epub 2020 Dec 17. PMID 33332778
- [Background] FDA. EMERGENCY USE AUTHORIZATION (EUA) OF REGEN-COV (casirivimab and imdevimab): Food and Drug Adminsteration (FDA); 2021 [updated 16/9/2021. first:[FACT SHEET FOR HEALTH CARE PROVIDERS,]. Available from: https://www.fda.gov/media/145611/download
- [Background] WHO COVID19 disease progression ordinal scale. February 18, 2020. [Available from: https://www.who.int/blueprint/priority-diseases/key-action/COVID-19_Treatment_Trial_Design_Master_Protocol_synopsis_Final_18022020.pdf
- [Background] Placais L, Richier Q, Noel N, Lacombe K, Mariette X, Hermine O. Immune interventions in COVID-19: a matter of time? Mucosal Immunol. 2022 Feb;15(2):198-210. doi: 10.1038/s41385-021-00464-w. Epub 2021 Oct 28. PMID 34711920
- [Background] Yang Z, Hu Q, Huang F, Xiong S, Sun Y. The prognostic value of the SOFA score in patients with COVID-19: A retrospective, observational study. Medicine (Baltimore). 2021 Aug 13;100(32):e26900. doi: 10.1097/MD.0000000000026900. PMID 34397917
- [Derived] Hegazy SK, Tharwat S, Hassan AH. Clinical study to compare the efficacy and safety of casirivimab & imdevimab, remdesivir, and favipravir in hospitalized COVID-19 patients. J Clin Virol Plus. 2023 Jun;3(2):100151. doi: 10.1016/j.jcvp.2023.100151. Epub 2023 May 10. PMID 37220480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from 1/11/2021 to 29/5/2022 at isolation hospital, Mansoura university
Pre-assignment Details: assignment is applied after admission of participants
Period: Overall Study
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Started | 53 | 106 | 106
Completed | 53 | 106 | 106
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir | Total
Number analyzed (Participants) | 53 | 106 | 106 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.34 (16.096) | 59.3 (15.98) | 65.02 (14.26) | 60.88 (15.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 42 | 61 | 127
  Male | 29 | 64 | 45 | 138
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Middle eastern | 53 | 106 | 106 | 265
Number of co-morbidities [Count of Participants; unit: Participants]
  0 | 10 | 32 | 22 | 64
  1 | 16 | 27 | 19 | 62
  2 | 14 | 28 | 33 | 75
  3 | 11 | 16 | 18 | 45
  4 | 2 | 2 | 10 | 14
  5 | 0 | 1 | 3 | 4
  6 | 0 | 0 | 1 | 1
Method of diagnosis [Count of Participants; unit: Participants]
  symptoms | 0 | 0 | 0 | 0
  laboratory and radiology | 0 | 0 | 0 | 0
  polymerase chain reaction confirmed | 53 | 106 | 106 | 265
Severity of COVID-19 [Count of Participants; unit: Participants]
  moderate | 18 | 20 | 20 | 58
  severe | 27 | 60 | 53 | 140
  critical | 8 | 26 | 33 | 67
World health organization clinical progression scale [Count of Participants; unit: Participants] — 0. Uninfected
  Ambulatory mild disease
  1. Asymptomatic; viral RNA detected
  2. Symptomatic; independent.
  3. Symptomatic; assistance needed
     Hospitalized: moderate disease
  4. Hospitalized; no oxygen therapy
  5. Hospitalized; oxygen by mask or nasal prongs
     Hospitalized: sever disease
  6. Hospitalized; oxygen by NIV or high flow
  7. Intubation and mechanical ventilation, pO2 /FIO2 ≥ 150 or Spo2 /FiO2 ≥200
  8. Mechanical ventilation pO2/FiO2 <150 (SpO2 /FiO2 < 200) or vasopressors
  9. Mechanical ventilation pO2 / FiO2 < 150 and vasopressors, dialysis or ECMO
     Dead
  10. Dead
  Participants
    3 | 0 | 1 | 0 | 1
    4 | 15 | 5 | 10 | 30
    5 | 35 | 100 | 96 | 231
    6 | 3 | 0 | 0 | 3
Number of symptoms [Count of Participants; unit: Participants]
  2 | 4 | 2 | 2 | 8
  3 | 13 | 6 | 4 | 23
  4 | 32 | 97 | 97 | 226
  5 | 4 | 1 | 3 | 8
Antibiotics use [Count of Participants; unit: Participants]
  yes | 53 | 106 | 106 | 265
  no | 0 | 0 | 0 | 0
macrolide use [Count of Participants; unit: Participants]
  yes | 8 | 8 | 2 | 18
  no | 45 | 98 | 104 | 247
fluoroquinolone use [Count of Participants; unit: Participants]
  yes | 41 | 92 | 95 | 228
  no | 12 | 14 | 11 | 37
cephalosporin use [Count of Participants; unit: Participants]
  yes | 39 | 86 | 83 | 208
  no | 14 | 20 | 23 | 57
carbapenem use [Count of Participants; unit: Participants]
  yes | 10 | 32 | 22 | 64
  no | 43 | 74 | 84 | 201
piperacillin use [Count of Participants; unit: Participants]
  yes | 0 | 0 | 0 | 0
  no | 53 | 106 | 106 | 265
amoxicillin/ clavulanate use [Count of Participants; unit: Participants]
  yes | 0 | 0 | 0 | 0
  no | 53 | 106 | 106 | 265
co-trimoxazole use [Count of Participants; unit: Participants]
  yes | 0 | 0 | 0 | 0
  no | 53 | 106 | 106 | 265
linezolide use [Count of Participants; unit: Participants]
  yes | 5 | 12 | 4 | 21
  no | 48 | 94 | 102 | 244
teicoplanin use [Count of Participants; unit: Participants]
  yes | 1 | 0 | 2 | 3
  no | 52 | 106 | 104 | 262
Anticoagulant use [Count of Participants; unit: Participants]
  yes | 49 | 101 | 96 | 246
  no | 4 | 5 | 10 | 19
dose of anticoagulant [Count of Participants; unit: Participants]
  prophylactic | 39 | 80 | 81 | 200
  therapeutic | 14 | 26 | 25 | 65
Antiplatelet use [Count of Participants; unit: Participants]
  yes | 5 | 6 | 0 | 11
  no | 48 | 100 | 106 | 254
Steriods use [Count of Participants; unit: Participants]
  yes | 45 | 105 | 98 | 248
  no | 8 | 1 | 8 | 17
Additive therapy use [Count of Participants; unit: Participants]
  yes | 51 | 106 | 105 | 262
  no | 2 | 0 | 1 | 3
paracetamol use [Count of Participants; unit: Participants]
  yes | 50 | 105 | 106 | 261
  no | 3 | 1 | 0 | 4
zinc use [Count of Participants; unit: Participants]
  yes | 4 | 0 | 1 | 5
  no | 49 | 106 | 105 | 260
acetylcysteine use [Count of Participants; unit: Participants]
  yes | 52 | 106 | 106 | 264
  no | 1 | 0 | 0 | 1
lactoferrin use [Count of Participants; unit: Participants]
  yes | 1 | 0 | 0 | 1
  no | 52 | 106 | 106 | 264
vitamin C use [Count of Participants; unit: Participants]
  yes | 4 | 7 | 1 | 12
  no | 49 | 99 | 105 | 253
Oxygen therapy use [Count of Participants; unit: Participants]
  yes | 37 | 99 | 102 | 238
  no | 16 | 7 | 4 | 27
Nasal Prongs use [Count of Participants; unit: Participants]
  yes | 18 | 35 | 39 | 92
  no | 35 | 71 | 67 | 173
Simple Face Mask use [Count of Participants; unit: Participants]
  yes | 30 | 82 | 87 | 199
  no | 23 | 24 | 19 | 66
Mask Reservoir use [Count of Participants; unit: Participants]
  yes | 8 | 33 | 14 | 55
  no | 45 | 73 | 92 | 210
High Flow Nasal Cannula use [Count of Participants; unit: Participants]
  yes | 5 | 22 | 18 | 45
  no | 48 | 84 | 88 | 220
Continuous Positive Attenuated Pressure use [Count of Participants; unit: Participants]
  yes | 4 | 39 | 36 | 79
  no | 49 | 67 | 70 | 186
Invasive Mechanical Ventilation use [Count of Participants; unit: Participants]
  yes | 1 | 29 | 29 | 59
  no | 52 | 77 | 77 | 206
Vasopressor use [Count of Participants; unit: Participants]
  yes | 0 | 23 | 18 | 41
  no | 53 | 83 | 88 | 224
Prone Positioning [Count of Participants; unit: Participants]
  yes | 0 | 5 | 9 | 14
  no | 53 | 101 | 97 | 251
Heart rate [Mean (Standard Deviation); unit: beats/ minute] | 82.40 (12.443) | 85.7 (16.072) | 87.02 (16.79) | 85.04 (15.1)
Respiratory rate [Mean (Standard Deviation); unit: breaths/ minute] | 24.25 (3.246) | 25.4 (5.58) | 24.72 (5.012) | 24.79 (4.612)
Body temperature [Mean (Standard Deviation); unit: degree Celsius] | 36.951 (0.492) | 36.938 (0.456) | 36.906 (1.18) | 36.92 (0.709)
O2 saturation on Oxygen therapy [Mean (Standard Deviation); unit: percentage of O2 saturation] | 96.26 (2.391) | 95.86 (3.795) | 96.01 (3.130) | 96.04 (3.105)
O2 saturation on Room air [Mean (Standard Deviation); unit: percentage of O2 saturation] | 92.36 (4.816) | 87.62 (7.171) | 88.35 (7.006) | 89.44 (6.33)
Aspartate aminotransferase level [Mean (Standard Deviation); unit: Units/liter] | 45.62 (38.619) | 52.95 (35.49) | 54.52 (67.85) | 51.03 (47.319)
Alanine aminotransferase level [Mean (Standard Deviation); unit: Units/liter] | 33.34 (27.166) | 33.27 (22.826) | 42.79 (77.37) | 36.46 (42.454)
Bilirubin level [Mean (Standard Deviation); unit: milligram/deciliter] | 0.5472 (0.299) | 0.6228 (0.79) | 0.7327 (0.69) | 0.634 (0.593)
Albumin level [Mean (Standard Deviation); unit: gram/deciliter] | 3.1774 (0.461) | 3.1715 (0.48) | 3.1021 (0.512) | 3.15 (0.484)
Prothrombin Time [Mean (Standard Deviation); unit: seconds] — the time it takes for the liquid portion (plasma) of your blood to clot.
  seconds | 14.575 (1.68) | 15.338 (1.997) | 15.69 (2.476) | 15.201 (2.051)
International normalized ratio [Mean (Standard Deviation); unit: Ratio] — a ratio of the patient's PT to a control PT standardized for the potency of the thromboplastin reagent developed by the World Health Organization (WHO) using the following formula: INR = Patient PT/ Control PT.
  normal value is 1 higher value means higher tendency for bleeding lower value means higher tendency for clotting
  Ratio | 1.2625 (0.201) | 1.3436 (0.239) | 1.3868 (0.296) | 1.33 (0.245)
Serum creatinine [Mean (Standard Deviation); unit: milligram/deciliter] | 1.2092 (1.355) | 1.0999 (0.924) | 1.8807 (1.912) | 1.3966 (1.397)
Total leukocytic count [Mean (Standard Deviation); unit: 10^3 cells/mm^3] | 8.6934 (4.129) | 8.4562 (5.044) | 11.0268 (9.4) | 9.39 (6.191)
Lymphocyte count [Mean (Standard Deviation); unit: 10^9 cells/L] | 0.9658 (0.521) | 0.9123 (0.429) | 1.4834 (5.62) | 1.12 (2.19)
Hemoglobin level [Mean (Standard Deviation); unit: gram/deciliter] | 12.59 (1.58) | 12.44 (2.07) | 11.94 (2.54) | 12.32 (2.063)
Hematocrit level [Mean (Standard Deviation); unit: percentage of total blood volume] | 39.317 (6.045) | 36.975 (5.586) | 35.259 (8.559) | 37.18 (6.73)
Platelet count [Mean (Standard Deviation); unit: 10^3 cells/uL] | 234.913 (91.5) | 211.613 (92.3) | 217.591 (122) | 221.37 (101.93)
Lactate dehydrogenase level [Mean (Standard Deviation); unit: international units per liter] | 413.06 (294.7) | 389.81 (222.668) | 378.5 (250.183) | 393.79 (255.85)
Creatine kinase level [Mean (Standard Deviation); unit: Units/liter] | 185.96 (207.6) | 228.07 (367.1) | 232.75 (287) | 215.59 (287.23)
D-dimer level [Mean (Standard Deviation); unit: μg/mL] | 0.6189 (0.493) | 0.1433 (0.227) | 0.2915 (0.385) | 0.351 (0.368)
C-reactive protein level [Mean (Standard Deviation); unit: milligram/liter] | 61.566 (39.71) | 61.292 (35.3) | 95.513 (157.8) | 72.79 (77.60)
Ferritin level [Mean (Standard Deviation); unit: micrograms per liter] | 442.34 (190.4) | 418.06 (193.8) | 1158.4 (6953) | 672.93 (2445.73)
Sodium level [Mean (Standard Deviation); unit: millimole/liter] | 146.472 (30.7) | 145.243 (20) | 144.315 (18.5) | 145.34 (23.06)
Potassium level [Mean (Standard Deviation); unit: millimole/liter] | 3.6228 (0.514) | 3.47 (0.674) | 3.79 (0.829) | 3.627 (0.672)
arterial oxygen pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 36.689 (12.59) | 37.325 (14.6) | 37.603 (12.08) | 37.205 (13.09)
ratio of arterial Oxygen pressure to fraction inspired of Oxygen [Mean (Standard Deviation); unit: Ratio] — PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage) also known as the Horowitz index, the Carrico index, and (most conveniently) the P/F ratio. The PaO2/FiO2 ratio is frequently used to determine the severity of lung injury in mechanically ventilated patients.
  normal >300 mild ARDS(acute respiratory distress syndrome)= 200-300 moderate ARDS= 100-200 severe ARDS <100
  Ratio | 223.5057 (207) | 156.7358 (171) | 164.142 (138) | 181.46 (516)
Glasgow coma score [Count of Participants; unit: Participants] — minimum 0 means dead maximum 15 means fully conscious higher score means better consciousness Eye opening response spontaneous 4 To verbal command 3 To pain 2 None 1 Verbal response Oriented conversation 5 Disoriented conversation 4
  Inappropriate words Incomprehensible words 3 Incomprehensible sound 2 None 1 Motor response Obeys verbal command 6 Localized painful stimuli 5 Flexion withdrawal from painful stimuli 4 Decorticate response to painful stimuli 3 None 1
  Participants
    4 | 0 | 2 | 0 | 2
    6 | 0 | 1 | 0 | 1
    8 | 0 | 0 | 1 | 1
    9 | 0 | 0 | 1 | 1
    10 | 0 | 2 | 8 | 10
    13 | 0 | 0 | 3 | 3
    14 | 1 | 4 | 7 | 12
    15 | 52 | 97 | 86 | 235
Sequential organ function assessment [Count of Participants; unit: Participants] — minimum 0 maximum 24 higher score means worse case PaO2/FiO2 0(> 400) 1(≤ 400) 2(≤ 300) 3(≤ 200 with respiratory support) 4(≤ 100 with respiratory support),Platelets 0 >150 1 101-150 2 51-100 3 21-50 4 ≤20, bilirubin 0 <1.2 mg/dl1 1.2-1.9 mg/dl 2 2-5.9 mg/dl 3 6-11.9 mg/dl 4 >12 mg/dl, Blood Pressure 0 no Hypotension 1MAP< 70 mmHg2 On dopamine≤ 5 mcg/Kg/min 3 On dopamine > 5 mcg/ kg/ min , 4 On dopamine >15 mcg/ kg/ min or epinephrine >0.1,GCS0 (15)1(13-14)2(10-12) 3(6-9) 4(<6), Renal function Creatinine 0 < 1.2 1 1.2-1.92 2-3.4 3 3.5-4.9 4 >5
  Participants
    0 | 11 | 2 | 1 | 14
    1 | 1 | 1 | 4 | 6
    2 | 3 | 9 | 3 | 15
    3 | 12 | 25 | 17 | 54
    4 | 17 | 36 | 28 | 81
    5 | 7 | 18 | 17 | 42
    6 | 0 | 6 | 13 | 19
    7 | 2 | 4 | 9 | 15
    8 | 0 | 3 | 7 | 10
    9 | 0 | 1 | 3 | 4
    10 | 0 | 1 | 3 | 4
    14 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 28-days Mortality Rate
Description: Dead or alive
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  dead | 1 | 34 | 43
  alive | 52 | 72 | 63
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.176, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

2. Primary Outcome: Number of Participants With Positive or Negative Polymerase Chain Reaction (PCR) Test Results at End of Hospital Visit
Description: positive or negative
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  positive | 36 | 92 | 78
  negative | 17 | 14 | 28
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.011, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.021, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.42, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.007, Kruskal-Wallis

3. Primary Outcome: Number of Participants With Infusion Related Reactions, Hypersensitivity Reactions and Any Serious Adverse Events
Description: yes or no
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  yes | 0 | 0 | 0
  no | 53 | 106 | 106
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.99, Kruskal-Wallis

4. Secondary Outcome: Need for Invasive Mechanical Ventilation
Description: yes or no
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  yes | 1 | 22 | 22
  no | 52 | 84 | 84
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.005, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.99, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.003, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.003, Kruskal-Wallis

5. Secondary Outcome: Oxygen Support Duration (Days)
Description: in days
Time Frame: up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
days | 3.72 (3.527) | 9.2 (7.107) | 7.46 (5.077)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.119, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

6. Secondary Outcome: Time to Clinical Improvement (Defined as 2 Points Reduction in the WHO Disease Ordinal Progression Scale or Discharge, Whatever Happens First
Description: in days
  WHO disease ordinal progression scale 0= Uninfected Ambulatory mild disease
  1. Asymptomatic; viral RNA detected
  2. Symptomatic; independent.
  3. Symptomatic; assistance needed Hospitalized: moderate disease
  4. Hospitalized; no oxygen therapy
  5. Hospitalized; oxygen by mask or nasal prongs Hospitalized: sever disease
  6. Hospitalized; oxygen by NIV or high flow
  7. Intubation and mechanical ventilation, pO2 /FIO2 ≥ 150 or Spo2 /FiO2 ≥200
  8. Mechanical ventilation pO2/FiO2 <150 (SpO2 /FiO2 < 200) or vasopressors
  9. Mechanical ventilation pO2 / FiO2 < 150 and vasopressors, dialysis or ECMO Dead
  10. Dead
Time Frame: up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
days | 7.4 (3.101) | 8.33 (6.38) | 7.75 (4.265)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.933, Kruskal-Wallis

7. Secondary Outcome: Duration of Hospitalization
Description: in days
Time Frame: up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
days | 8.94 (3.165) | 11.85 (6.264) | 10.59 (5.26)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.011, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.054, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.185, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.004, Kruskal-Wallis

8. Secondary Outcome: Sequential Organ Function Assessment (SOFA) Score on Day 3
Description: minimum 0 to maximum 24, higher scores mean worse outcomes Platelets, ×10³/µL
  ≥150 0 100-149+1 50-99+2 20-49+3 <20+4
  Glasgow Coma Scale If on sedatives, estimate assumed GCS off sedatives 15 0 13-14+1 10-12+2 6-9+3 <6+4
  Bilirubin, mg/dL (μmol/L) <1.2 (<20) 0 1.2-1.9 (20-32)+1 2.0-5.9 (33-101)+2 6.0-11.9 (102-204)+3 ≥12.0 (>204)+4
  Mean arterial pressure OR administration of vasoactive agents required Listed doses are in units of mcg/kg/min No hypotension 0 MAP <70 mmHg+1 DOPamine ≤5 or DOBUTamine (any dose)+2 DOPamine >5, EPINEPHrine ≤0.1, or norEPINEPHrine ≤0.1+3 DOPamine >15, EPINEPHrine >0.1, or norEPINEPHrine >0.1+4
  Creatinine, mg/dL (μmol/L) (or urine output) <1.2 (<110) 0 1.2-1.9 (110-170)+1 2.0-3.4 (171-299)+2 3.5-4.9 (300-440) or UOP <500 mL/day+3
  ≥5.0 (>440) or UOP <200 mL/day+4
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  0 | 12 | 1 | 1
  1 | 3 | 8 | 6
  2 | 12 | 12 | 8
  3 | 18 | 24 | 16
  4 | 6 | 40 | 18
  5 | 0 | 4 | 16
  6 | 0 | 5 | 11
  7 | 1 | 4 | 12
  8 | 0 | 4 | 3
  9 | 1 | 1 | 7
  10 | 0 | 0 | 1
  11 | 0 | 0 | 3
  12 | 0 | 2 | 1
  13 | 0 | 1 | 2
  16 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.001, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

9. Secondary Outcome: COVID-19 World Health Organization (WHO) Disease Progression Scale at Day 3
Description: minimum 0 to maximum 10, higher scores mean worse outcomes
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 52 | 106 | 106
Participants
  WHO scale 3 | 0 | 1 | 0
  WHO scale 4 | 25 | 17 | 17
  WHO scale 5 | 20 | 57 | 58
  WHO scale 6 | 7 | 28 | 22
  WHO scale 8 | 0 | 0 | 5
  WHO scale 9 | 0 | 2 | 4
  WHO scale 10 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.758, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

10. Secondary Outcome: Aspartate Aminotransferase (AST) at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Units/liter | 48.53 (60.487) | 48.67 (41.128) | 43.93 (36.497)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.412, Kruskal-Wallis

11. Secondary Outcome: Ferritin at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
micrograms per liter | 393.04 (170.2) | 427.25 (194.8) | 1110 (6784.6)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.106, Kruskal-Wallis

12. Secondary Outcome: Lactate Dehydrogenase (LDH) at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: international units per liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
international units per liter | 351.27 (258.57) | 404.45 (214.92) | 354.7 (204.2)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.01, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.06, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.156, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.003, Kruskal-Wallis

13. Secondary Outcome: D-dimer at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
μg/mL | 0.244 (0.2211) | 0.23 (0.3321) | 0.29 (0.3845)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.219, Kruskal-Wallis

14. Secondary Outcome: Alanine Aminotransferase (ALT) at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Units/liter | 33.62 (34.535) | 36.46 (32.585) | 36.16 (49.86)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.298, Kruskal-Wallis

15. Secondary Outcome: Albumin at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: gm/dl
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
gm/dl | 3.157 (0.3858) | 2.947 (0.4507) | 2.854 (0.504)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.015, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.232, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.004, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.054, Kruskal-Wallis

16. Secondary Outcome: Bilirubin at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
milligram/deciliter | 0.4793 (0.255) | 0.6457 (0.654) | 0.7053 (0.86)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.68, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.232, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.004, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.054, Kruskal-Wallis

17. Secondary Outcome: C-reactive Protein (CRP) at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: milligram/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 52 | 106 | 82
milligram/liter | 33.89 (31.44) | 52.61 (37.719) | 64.1 (63.035)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.002, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.557, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.004, Kruskal-Wallis

18. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Description: duration of ICU stay
Time Frame: up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
days | 1.45 (1.835) | 7.6 (7.614) | 6.69 (6.23)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.51, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

19. Secondary Outcome: C-reactive Protein (CRP) at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: milligram/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
milligram/liter | 14.06 (14.548) | 47.43 (52.631) | 65.73 (90.34)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.891, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

20. Secondary Outcome: C-reactive Protein (CRP) at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: milligram/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
milligram/liter | 7.5 (5.745) | 37.05 (55.395) | 39.31 (54.77)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.516, Kruskal-Wallis

21. Secondary Outcome: C-reactive Protein (CRP) at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: milligram/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
milligram/liter |  | 39 (38.419) | 96 (NA) — The number of participants is 1, so the Standard Deviation was not calculated
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.264, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Sequential Organ Function Assessment (SOFA) Score on Day 7
Description: minimum 0 to maximum 24, higher scores mean worse outcomes
Time Frame: day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
Participants
  0 | 5 | 1 | 1
  1 | 18 | 4 | 4
  2 | 12 | 10 | 10
  3 | 3 | 13 | 13
  4 | 0 | 28 | 7
  5 | 1 | 7 | 7
  6 | 0 | 6 | 5
  7 | 0 | 2 | 6
  8 | 0 | 1 | 4
  9 | 0 | 2 | 2
  10 | 0 | 4 | 2
  11 | 0 | 3 | 3
  12 | 0 | 0 | 3
  13 | 0 | 1 | 2
  14 | 0 | 1 | 2
  15 | 0 | 1 | 2
  16 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.256, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

23. Secondary Outcome: Sequential Organ Function Assessment Score (SOFA) on Day 14
Description: minimum 0 to maximum 24, higher scores mean worse outcomes
Time Frame: day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 16
Participants
  0 | 3 | 1 | 0
  1 | 1 | 1 | 1
  2 | 0 | 1 | 1
  3 | 0 | 2 | 3
  4 | 0 | 4 | 3
  5 | 0 | 4 | 2
  6 | 0 | 0 | 1
  8 | 0 | 2 | 2
  9 | 0 | 1 | 1
  11 | 0 | 2 | 0
  12 | 0 | 0 | 1
  14 | 0 | 1 | 0
  16 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.008, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.797, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.003, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.004, Kruskal-Wallis

24. Secondary Outcome: Sequential Organ Function Assessment Score (SOFA) on Day 28
Description: minimum 0 to maximum 24, higher scores mean worse outcomes
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
Participants
  0 |  | 1 | 0
  3 |  | 1 | 0
  12 |  | 1 | 0
  13 |  | 1 | 0
  17 |  | 0 | 1
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.157, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: COVID-19 World Health Organization (WHO) Disease Progression Scale at Day 7
Description: minimum 0 to maximum 10, higher scores mean worse outcomes
Time Frame: day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
Participants
  4 | 28 | 20 | 21
  5 | 11 | 28 | 22
  6 | 0 | 26 | 16
  8 | 0 | 3 | 5
  9 | 0 | 7 | 4
  10 | 0 | 0 | 6
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.982, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

26. Secondary Outcome: COVID-19 World Health Organization (WHO) Disease Progression Scale at Day 14
Description: minimum 0 to maximum 10, higher scores mean worse outcomes
Time Frame: day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 16
Participants
  4 | 4 | 2 | 7
  5 | 0 | 8 | 4
  6 | 0 | 3 | 1
  8 | 0 | 3 | 1
  9 | 0 | 3 | 3
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.015, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.136, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.062, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.005, Kruskal-Wallis

27. Secondary Outcome: COVID-19 World Health Organization (WHO) Disease Progression Scale at Day 28
Description: minimum 0 to maximum 10, higher scores mean worse outcomes
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
Participants
  5 |  | 2 | 0
  9 |  | 2 | 0
  10 |  | 0 | 1
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.136, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Aspartate Aminotransferase (AST) at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
Units/liter | 41.77 (32.465) | 35.26 (20.089) | 41.35 (39.78)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.687, Kruskal-Wallis

29. Secondary Outcome: Aspartate Aminotransferase (AST) at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
Units/liter | 26.75 (18.118) | 22.79 (13.319) | 30.19 (16.802)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.278, Kruskal-Wallis

30. Secondary Outcome: Aspartate Aminotransferase (AST) at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
Units/liter |  | 31 (11.605) | 27 (NA) — The number of participants is 1, so the Standard Deviation was not calculated
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Alanine Aminotransferase (ALT) at Day 7
Description: Continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
Units/liter | 26 (18.604) | 30.54 (23.062) | 33.90 (33.58)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.574, Kruskal-Wallis

32. Secondary Outcome: Alanine Aminotransferase (ALT) at Day 14
Description: Continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
Units/liter | 15.75 (4.856) | 22.42 (15.788) | 35.38 (17.55)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.017, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.017, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.041, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.616, Kruskal-Wallis

33. Secondary Outcome: Alanine Aminotransferase (ALT) at Day 28
Description: Continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
Units/liter |  | 71.75 (57) | 39.5 (NA) — The number of participants is 1, so the Standard Deviation was not calculated
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.99, Kruskal-Wallis

34. Secondary Outcome: Bilirubin at Day 7
Description: Continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
milligram/deciliter | 0.3717 (0.221) | 0.6575 (0.699) | 0.8886 (1.54)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.208, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.001, Kruskal-Wallis

35. Secondary Outcome: Bilirubin at Day 14
Description: Continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
milligram/deciliter | 0.3625 (0.11) | 0.494 (0.2229) | 0.6888 (0.37)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.088, Kruskal-Wallis

36. Secondary Outcome: Bilirubin at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
milligram/deciliter |  | 0.41 (0.14376) | 1.67 (NA) — The number of participants is 1, so the Standard Deviation was not calculated
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.157, Wilcoxon (Mann-Whitney)

37. Secondary Outcome: Albumin at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: gm/dl
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
gm/dl | 2.98 (0.4073) | 2.77 (0.4837) | 2.644 (0.489)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.006, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.151, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.035, Kruskal-Wallis

38. Secondary Outcome: Albumin at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: gm/dl
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
gm/dl | 3.425 (0.2872) | 2.82 (0.4184) | 2.813 (0.368)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.037, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.997, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.016, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.014, Kruskal-Wallis

39. Secondary Outcome: Albumin at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: gm/dl
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
gm/dl |  | 2.575 (0.3304) | 2.7 (NA) — The number of participants is 1, so the Standard Deviation was not calculated
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

40. Secondary Outcome: Platelets at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
10^3 cells/uL | 271.64 (97.62) | 253.425 (105) | 226.35 (116.2)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.047, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.04, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.036, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.67, Kruskal-Wallis

41. Secondary Outcome: Platelets at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
10^3 cells/uL | 268.829 (93.9) | 243.514 (116.2) | 212.76 (123.2)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.015, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.027, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.008, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.38, Kruskal-Wallis

42. Secondary Outcome: Platelets at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
10^3 cells/uL | 248 (136.48) | 216.95 (126.3) | 215.63 (126.3)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.814, Kruskal-Wallis

43. Secondary Outcome: Platelets at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
10^3 cells/uL |  | 246.75 (113) | 15 (NA) — Standard Deviation not calculable as only 1 participant was analyzed
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.157, Wilcoxon (Mann-Whitney)

44. Secondary Outcome: Serum Creatinine (S.Cr) at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
milligram/deciliter | 1.0769 (0.941) | 0.9546 (0.865) | 1.6568 (1.776)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.971, Kruskal-Wallis

45. Secondary Outcome: Serum Creatinine (S.Cr) at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
milligram/deciliter | 0.9674 (0.752) | 0.9952 (0.987) | 1.6541 (1.9)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis

46. Secondary Outcome: Serum Creatinine (S.Cr) at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
milligram/deciliter | 0.775 (0.221) | 0.6316 (0.152) | 1.45 (1.7753)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.007, Kruskal-Wallis
Statistical Analysis 2: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.017, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.452, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.237, Kruskal-Wallis

47. Secondary Outcome: Serum Creatinine (S.Cr) at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
milligram/deciliter |  | 0.525 (0.1708) | 1.2 (NA) — Standard Deviation not calculable as only 1 participant was analyzed
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.157, Wilcoxon (Mann-Whitney)

48. Secondary Outcome: D-dimer at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
μg/mL | 0.109 (0.1483) | 0.319 (0.5017) | 0.425 (0.5678)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.015, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.223, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.004, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.05, Kruskal-Wallis

49. Secondary Outcome: D-dimer at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
μg/mL | 0.05 (0.1) | 0.41 (0.5999) | 0.313 (0.461)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.423, Kruskal-Wallis

50. Secondary Outcome: D-dimer at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
μg/mL |  | 0.4 (0.8) | 0.4 (NA) — Standard Deviation not calculable as only 1 participant was analyzed
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.429, Wilcoxon (Mann-Whitney)

51. Secondary Outcome: Creatine Kinase (Ck) at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Units/liter | 142.2 (135.12) | 197.94 (342.1) | 181.45 (166)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.089, Kruskal-Wallis

52. Secondary Outcome: Creatine Kinase (Ck) at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
Units/liter | 126.743 (112) | 211.9 (420.23) | 175.99 (155)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.222, Kruskal-Wallis

53. Secondary Outcome: Creatine Kinase (Ck) at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
Units/liter | 49.5 (30.116) | 122.89 (93.259) | 142.75 (176)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.252, Kruskal-Wallis

54. Secondary Outcome: Creatine Kinase (Ck) at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
Units/liter |  | 119.22 (88.21) | 134.25 (NA) — Standard Deviation not calculable as only 1 participant was analyzed
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.157, Wilcoxon (Mann-Whitney)

55. Secondary Outcome: Lactate Dehydrogenase (LDH) at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: international units per liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
international units per liter | 271.4 (165.99) | 371.37 (196.2) | 349.68 (201)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.007, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.382, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.017, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.002, Kruskal-Wallis

56. Secondary Outcome: Lactate Dehydrogenase (LDH) at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: international units per liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
international units per liter | 379.75 (313.9) | 360.89 (244.8) | 306.88 (266)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.457, Kruskal-Wallis

57. Secondary Outcome: Lactate Dehydrogenase (LDH) at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: international units per liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
international units per liter |  | 314.5 (108.99) | 270 (NA) — Standard Deviation not calculable as only 1 participant was analyzed
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

58. Secondary Outcome: Ferritin at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
micrograms per liter | 368.42 (167.8) | 450.37 (247.6) | 1433 (8174)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.01, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.605, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.003, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.01, Kruskal-Wallis

59. Secondary Outcome: Ferritin at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
micrograms per liter | 398.5 (131.43) | 637.37 (436) | 519.88 (431)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.293, Kruskal-Wallis

60. Secondary Outcome: Ferritin at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
micrograms per liter |  | 1355 (896.3) | 410 (NA) — Standard Deviation not calculable as only 1 participant was analyzed
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.157, Wilcoxon (Mann-Whitney)

61. Secondary Outcome: Incidence of Acute Kidney Injury (AKI)
Description: Incidence of acute kidney injury (AKI)
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  yes | 1 | 4 | 7
  no | 52 | 102 | 99
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.36, Kruskal-Wallis

62. Secondary Outcome: Incidence of Acute Liver Damage (ALD)
Description: Incidence of acute liver damage (ALD)
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  yes | 1 | 6 | 3
  no | 52 | 100 | 103
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.404, Kruskal-Wallis

63. Secondary Outcome: Day of Death
Description: day of death
Time Frame: up to 60 days
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
day | 0.19 (1.061) | 12.57 (6.22) | 10.13 (6.530)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.234, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

64. Secondary Outcome: Mortality at Discharge
Description: mortality at discharge
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  dead | 1 | 33 | 41
  alive | 52 | 73 | 65
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.223, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

65. Other Pre Specified Outcome: Glasgow Coma Score (GCS) at Day 3
Description: minimum 0 to maximum 15, higher scores mean better outcomes
Time Frame: day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Participants
  3 | 0 | 3 | 6
  4 | 0 | 1 | 0
  6 | 0 | 1 | 0
  7 | 0 | 0 | 1
  8 | 0 | 0 | 1
  9 | 0 | 0 | 1
  10 | 0 | 2 | 10
  12 | 0 | 0 | 1
  13 | 1 | 0 | 3
  14 | 1 | 5 | 6
  15 | 51 | 94 | 77
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.002, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.213, Kruskal-Wallis

66. Other Pre Specified Outcome: Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) at Day 3
Description: continuous level
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 53 | 106 | 106
Ratio | 298.57 (211.3) | 154.14 (138.9) | 166.96 (130)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.478, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

67. Other Pre Specified Outcome: Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) at Day 7
Description: continuous level
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
Ratio | 320.62 (93.64) | 163.55 (172.6) | 178.59 (138)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.413, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p < 0.001, Kruskal-Wallis

68. Other Pre Specified Outcome: Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) at Day 14
Description: continuous level
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
Ratio | 389.75 (51.93) | 154.67 (174) | 165.2 (98.87)
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.005, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.155, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p = 0.022, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.001, Kruskal-Wallis

69. Other Pre Specified Outcome: Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) at Day 28
Description: continuous level
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
Ratio |  | 172.75 (181) | 53 (NA) — Standard Deviation not calculable as only 1 participant was analyzed
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

70. Other Pre Specified Outcome: Glasgow Coma Score (GCS) at Day 7
Description: minimum 0 to maximum 15, higher scores mean better outcomes
Time Frame: day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 39 | 84 | 74
Participants
  3 | 0 | 10 | 13
  6 | 0 | 1 | 1
  7 | 0 | 0 | 1
  9 | 0 | 0 | 1
  10 | 0 | 3 | 11
  12 | 0 | 0 | 1
  13 | 0 | 1 | 1
  14 | 0 | 3 | 3
  15 | 39 | 66 | 42
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.003, Kruskal-Wallis
Statistical Analysis 3: Comparison: Casirivimab and Imdevimab vs Favipravir; Test type: Superiority; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Casirivimab and Imdevimab vs Remdesivir; Test type: Superiority; p = 0.011, Kruskal-Wallis

71. Other Pre Specified Outcome: Glasgow Coma Score (GCS) at Day 14
Description: minimum 0 to maximum 15, higher scores mean better outcomes
Time Frame: day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 4 | 19 | 13
Participants
  3 | 0 | 6 | 4
  10 | 0 | 0 | 0
  13 | 0 | 1 | 0
  14 | 0 | 1 | 2
  15 | 4 | 11 | 7
Statistical Analysis 1: Comparison: Casirivimab and Imdevimab vs Remdesivir vs Favipravir; Test type: Superiority; p = 0.189, Kruskal-Wallis

72. Other Pre Specified Outcome: Glasgow Coma Score (GCS) at Day 28
Description: minimum 0 to maximum 15, higher scores mean better outcomes
Time Frame: day 28
Population: patients who received casirivimab and imdevimab, not stayed at hospital until day of 28
Measure: Count of Participants; unit: Participants
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
Number analyzed (Participants) | 0 | 4 | 1
Participants
  3 |  | 2 | 1
  15 |  | 2 | NA — Standard Deviation not calculable as only 1 participant was analyzed
Statistical Analysis 1: Comparison: Remdesivir vs Favipravir; Test type: Superiority; p = 0.414, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: up to 60 days
Groups:
- Favipravir: Favipravir, tablets Day 1 (loading dose): 1600 mg (8 tablets) orally or in Ryle tube / 12 hours day 2-10 (maintenance dose): 800 mg (4 tablets) orally or in Ryle tube / 12 hours
  Favipiravir: antiviral drug
Arm/Group | Casirivimab and Imdevimab | Remdesivir | Favipravir
All-Cause Mortality (participants affected / at risk) | 1/53 | 34/106 | 43/106
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/106 | 0/106
Other Adverse Events (participants affected / at risk) | 0/53 | 0/106 | 0/106

LIMITATIONS AND CAVEATS:
1. applicable only on hospitalized COVID-19 patients (not include outpatients),
2. non-randomization of antiviral drugs among included patients,
3. non-blinding of interventions to investigators

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT05502081/Prot_SAP_ICF_002.pdf